CLINICAL TRIAL: NCT00463489
Title: Lifestyle Intervention Study in Adjuvant Treatment of Early Breast Cancer
Acronym: LISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OCOG-2007-LISA
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: lifestyle intervention; breast; cancer; adjuvant; letrozole; weight loss; BMI; post-menopausal; estrogen receptor positive; progesterone receptor positive
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mail-based (Active Comparator): Participants will receive a standardized mail-based intervention focussing on healthy living. This will include mailings at study entry as well as a two year subscription to health magazine.
  Interventions: Behavioral: Mail-based
- Individualized Lifestyle Intervention (Experimental): Women randomized to the individualized lifestyle intervention arm will receive an intervention program that consists of individual weight loss, diet and physical activity goals, incorporated into a 2 year standardized, structured telephone and mail-based intervention. In addition to diet and physical activity, the intervention will address behavioural and motivational issues relating to weight management including maintaining motivation, overcoming obstacles to success, relapse prevention, emotional distress, stress and time management.
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Women randomized to the lifestyle intervention arm will receive an intervention program that consists of individual weight loss, diet and physical activity goals, incorporated into a 2 year standardized, structured telephone and mail-based intervention. In addition to diet and physical activity, the intervention will address behavioural and motivational issues relating to weight management including maintaining motivation, overcoming obstacles to success, relapse prevention, emotional distress, stress and time management.
  Arms: Individualized Lifestyle Intervention
Behavioral: Mail-based — Participants will receive a standardized mail-based intervention focussing on healthy living. This will include mailings at study entry as well as a two year subscription to health magazine.
  Arms: Mail-based

SUMMARY:
The primary objective of this trial is to evaluate the effect of the addition of a 2 year, centrally delivered individualized, telephone-based lifestyle intervention focusing on weight management to a mailed educational intervention on Disease Free Survival in post-menopausal women with early stage breast cancer (hormone receptor positive), BMI ≥24-<40 kg/m2, who are receiving standard letrozole adjuvant therapy.

DETAILED DESCRIPTION:
The primary objective of this trial is to evaluate the effect of the addition of a 2 year, centrally delivered individualized, telephone-based lifestyle intervention focusing on weight management to a mailed educational intervention on Disease Free Survival in post-menopausal women with early stage breast cancer (hormone receptor positive), BMI ≥24-<40 kg/m2, who are receiving standard letrozole adjuvant therapy. The telephone intervention will involve 19 phone calls, as well as mailings and a participant manual; women will be asked to lose up to 10% of their weight by reducing their caloric and fat intake (by 500-1000 kcal/day, 20% calories fat) and increasing their moderate physical activity (to 150-200 minutes/week). Secondary outcomes include overall survival, distant disease-free survival, weight change, health-related quality of life (HRQOL), selected non-cancer medical events and biologic factors (notably insulin). Approximately 2,150 women will be enrolled; follow-up will continue until target event rates have been met (anticipated 4-6 years after completion of the intervention). This sample size will provide 80% power (type 1 error 0.05 2-tailed) to detect a hazard ratio (HR) for DFS of 0.74-0.76 in the weight loss intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal woman with a diagnosis of invasive breast cancer (T1-3,pN0-2,M0) for which definitive surgery was performed during the previous 36 months.
* On adjuvant hormonal therapy with letrozole at time of randomization (either as initial adjuvant hormonal therapy or after a switch from tamoxifen or other hormonal therapy).
* BMI ≥ 24 kg/m2.
* Medical, surgical or radiation oncologist agrees to subject participation in a diet and physical activity program.

Exclusion Criteria:

* Life expectancy less than five years.
* Self-reported inability to walk at least 2 blocks (at any pace).
* Insulin requiring diabetes (telephone directed diet and physical activity changes would be difficult in this population without close coordination with the treating physician). Non-insulin requiring diabetics are eligible for the study.
* Serious digestive and/or absorptive problems, including inflammatory bowel disease and chronic diarrhea that preclude adherence to the study diet.
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity. Moderate arthritis that does not preclude physical activity is not a reason for ineligibility.
* Psychiatric disorders or conditions that, in the opinion of the investigator, would preclude participation in the study intervention (e.g. untreated major depression or psychosis, substance abuse, severe personality disorder).
* Patients on aromatase inhibitors other than letrozole at study entry.
* Known recurrence of breast cancer (local, regional or distant) at any time prior to study entry.
* History of other malignancies except: adequately treated non-melanoma skin cancer, curatively treated in situ carcinoma of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years. Prior in situ cancer of the breast is not a reason for exclusion.
* Patients not fluent in either English or French (spoken and written).
* Patient unwilling or unable to provide informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2007-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 8 years

SECONDARY OUTCOMES:
Overall survival | 8 years
Distant disease-free survival | 8 years
Weight at 6, 12, 24, 36, 48 and 60 months compared to baseline | 5 years
Health-related quality of life at 6, 12, 24, 36, 48 and 60 months compared to baseline | 5 years
Other medical endpoints such as diabetes, cardiovascular disease, arthritis, fasting biomarkers at 12 months compared to baseline (for women participating in a biospecimen substudy) | 8 years
Compliance with study procedures. | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Goodwin, MD, MSc, Principal Investigator — UHN-Mount Sinai Hospital, Toronto, ON
Locations (21):
- United States (4):
  - Los Angeles Biomedical (LABIOMED) Research Institue at Harbor-UCLA Medical Center, Torrance, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Centre, Boston, Massachusetts
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (17):
  - Bcca - Csi, Kelowna, British Columbia
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Grand River Regional Cancer Centere, Kitchener, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Scarborough Hospital, Scarborough Village, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Trillium Healthcare Centre, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - CHUM - Hotel Dieu de Montreal, Montreal, Quebec

REFERENCES:
- [Background] Goodwin PJ, Segal RJ, Vallis M, Ligibel JA, Pond GR, Robidoux A, Blackburn GL, Findlay B, Gralow JR, Mukherjee S, Levine M, Pritchard KI. Randomized trial of a telephone-based weight loss intervention in postmenopausal women with breast cancer receiving letrozole: the LISA trial. J Clin Oncol. 2014 Jul 20;32(21):2231-9. doi: 10.1200/JCO.2013.53.1517. Epub 2014 Jun 16. PMID 24934783